CLINICAL TRIAL: NCT04468048
Title: Music Utilization in Sedation and Induction in Colonoscopy
Acronym: MUSIC
Status: Withdrawn | Type: Observational
Why Stopped: No participants
Sponsor: The Brooklyn Hospital Center (Other)
Responsible Party: Sponsor
Other Study IDs: 1309407-1
Record Dates: First submitted 2019-01-15; First posted 2020-07-13 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Colonoscopy
Keywords: Colonoscopy; Music; Propofol; Conscious Sedation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Music: Subjects will put on headphones containing music from the album "Nada Himalaya" performed by S. G. Sachchidananda. The music will start playing 10 minutes before the colonoscopy procedure and will stop once subjects have woken up from sedation. Subjects will be instructed to not tell anyone if music is playing from their headphones. Subjects will two questionnaires before the procedure asking about their initial anxiety levels and previous procedure history. Two questionnaires following the procedure will be provide asking about their anxiety levels following the procedure and their overall satisfaction with the procedure.
  Interventions: Other: Music: "Nada Himalaya" performed by S. G. Sachchidananda
- Control: Subjects will put on headphones, but there will be no music playing. Subjects are instructed to not tell anyone if music is playing from their headphones. Subjects will two questionnaires before the procedure asking about their initial anxiety levels and previous procedure history. Two questionnaires following the procedure will be provide asking about their anxiety levels following the procedure and their overall satisfaction with the procedure.

INTERVENTIONS:
Other: Music: "Nada Himalaya" performed by S. G. Sachchidananda — Music: "Nada Himalaya" performed by S. G. Sachchidananda
  Groups: Music

SUMMARY:
Conscious sedation (CS) if often used in the field of gastroenterology to alleviate pain and discomfort with interventional procedures. Although CS is relatively safe, there is concern for the development of cardiopulmonary complications. Music has been shown in multiple studies to decrease anxiety and improve patient satisfaction following cardiac, pulmonary, and surgical procedures. This is a prospective single-blinded randomized control trial that will examine the effects of active music participation and music listening on patients undergoing colonoscopy through propofol use (monitored anesthesia) at The Brooklyn Hospital Center. The study will enroll patients who will undergo colonoscopy from November 2018 to April 2019 and randomize them to receive music or no music starting at the initial nursing evaluation in the pre-procedure area. We hypothesize that incorporating music during colonoscopy procedures will alleviate patient discomfort, reduce narcotic/sedative usage and post-operative complications.

DETAILED DESCRIPTION:
Introduction Conscious sedation (CS) in the field of gastroenterology is commonly incorporated in order to alleviate pain and discomfort associated with interventional procedures. The use of CS to combat patient anxiety has been well documented [1]. Although CS is relatively safe, it is not immune to cardiopulmonary complications. Multiple studies have demonstrated a clear correlation between advancing age and procedure related complications [2-4]. It is also important to note that despite the lack of association between age and additional complications in a study conducted by Clarke et al, a third of their patients did not receive sedation/narcotic medications [5].

Obesity, which affects approximately two third of the U.S. population, has a myriad of health related risks and has been shown to contribute to the overall complications associated with endoscopic procedures [6]. Because those who are obese and overweight have higher than normal BMIs, BMI should not be ignored when assessing cardiopulmonary complications in patients undergoing endoscopic procedures. Moreover, a study by Qadeer et al. revealed that patients with high BMIs were more likely to experience hypoxic episodes [3].

A study by Sharma et al. (2007) looked at more than 300,000 patients who underwent endoscopic procedures while monitoring their risk factors for cardiopulmonary complications [4]. Older age, American Society of Anesthesia (ASA) grade value >2, inpatient procedures, and involvement of trainee with procedure were all shown to be associated with cardiopulmonary complications. In addition, another study by Bini et al.(2003) illustrated that the age of a patient, comorbid conditions, month of procedure (July and August), and midazolam dose were linked with increased negative outcomes [2]. The correlation between complication rate during procedures along with the year of the trainee conducting the procedure indirectly demonstrated the complications in the new academic year (July and August). Understanding that sedation during endoscopic procedures incurs significant risks particularly in patients who are underweight, obese or have numerous comorbidities can lead to steps aimed at better managing the aforementioned risks and reducing patient discomfort.

Music has been shown in many studies to decrease anxiety and improve patient satisfaction during and after procedures in cardiac, pulmonary and surgical procedures [7-16]. In regards to endoscopies, one hundred and eighty patients who were listening to music prior to endoscopic procedure had a significant reduction in stress compared to controls [17]. A similar type of study performed by Hayes et al. (year) revealed that music resulted in a statistically significant decrease in the State-Trait Anxiety Index (STAI) levels of patients undergoing an endoscopy [18] . In another study, music was played prior to and during procedure with no sedative/narcotic medications [19] . Patients with music experienced a decrease in blood pressure (BP) and RR compared to their counterparts who did not listen to music. A 3 point attitude scale showed that patients with music had less discomfort, illustrating that music has the potential to modulate physiological parameters. An instrumental composition from the album "Nada Himalaya" performed by S.G. Sachchidananda, was previously studied by Phanishree et al. (unpublished data), which demonstrated a decrease in the blood pressure and heart rate in patients. Furthermore, the patients were much more relaxed and calm compared to the beginning of the study. Other music genres have relaxation properties as well but we wanted to test one specific type of music to see proof of concept in colonoscopy before we introduce other genres.

Propofol is currently being used more frequently for the use of monitored anesthesia in surgical settings. Patients on propofol have a better recall that music was being played compared to general anesthesia, but they could not adequately recall the type of music [20]. Ambient room noise seems to be one of the main factors associated with increasing propofol requirements in an operation room (OR) which music seems to alleviate [21] . This has been further illustrated by the use of Bispectral index (BIS), which demonstrated increasing brain activity when OR decibels were over 50 [22]. With the initiation of music and propofol in the setting of spinal anesthesia, there was a significant decrease in propofol dose and cortisol levels intra-op demonstrating the stress relieving effect of music [23,24].

To fully monitor the sedation requirements for patients undergoing colonoscopy two different scales will be utilized to assess the depth of sedation. The validated University of Michigan Sedation Scale (UMSS) is a combination of auditory and visual stimuli that are used to assess the depth of sedation. Since Auditory stimuli can be difficult to assess with the headphones we will also utilize the Bispectral Index (BIS) to assess the depth of sedation. The BIS monitor is attached to an electrode that is fixed on the forehead of the patient and continually assesses the brain activity of the patient. A computer algorithm will assess the brain activity and gives a value that determines the level of sedation. This in conjunction with the UMSS scale will give an adequate representation of the depth of sedation. The UMSS is the standard of care (SOC) in colonoscopy and BIS in general anesthesia.

The UMSS scale:

0 - Awake and alert

1. - Minimally sedated: tired/sleepy, appropriate response to verbal conversation and/or sound
2. - Moderately sedated: somnolent/sleeping, easily aroused with light tactile stimulation or a simple verbal command
3. - Deeply sedated: deep sleep, arousable only with significant physical stimulation
4. - Unarousable

The initial propofol induction dosage is determined by the anesthesiologist and is given according to the mg/kg requirements. After the induction process the UMSS and BIS scores will be utilized to determine the amount of propofol to be given as IV pushes to achieve adequate sedation. Furthermore, the anesthesiologist routinely assesses the American society of Anesthesiology (ASA) grading system to determine the degree of risk associated with a procedure with each patient.

The ASA grading system:

Grade 1 Healthy person. Grade 2 Mild systemic disease. Grade 3 Severe systemic disease. Grade 4 Severe systemic disease that is a constant threat to life. Grade 5 A moribund person who is not expected to survive without the operation. Grade 6 A declared brain dead person whose organs are being removed for donor purposes.

Research Goals and Objectives This is a prospective single-blinded randomized controlled trial that will examine the effects of active music participation and music listening on patients undergoing colonoscopy via propofol (monitored anesthesia) at the Brooklyn Hospital Center. Our study aims to enroll patients who will undergo colonoscopy and randomize them to receive either music or no music starting at the time of initial nursing evaluation in the pre-procedure area. The primary endpoint is to assess the utilization of narcotics/sedatives during colonoscopy. Secondary endpoints include willingness to repeat the procedure, anxiety associated with procedure, and association between the year of trainee and the amount of narcotic/sedatives used in each arm of the study. The complications that occur in reference of the year of trainee will be observe. We hypothesize that incorporating music during colonoscopy procedures will alleviate patient discomfort, reduce narcotic/sedative usage and post-operative complications.

Study Design and Methodology

Design The study design chosen for this study is a prospective single-blinded randomized control trial as there will be a control group who will not be listening to music and treatment group. The period study will be conducted for the period of one year.

Study population The study population will include all individuals undergoing colonoscopies that consented to participating in the study. The study subjects will include the patients undergoing the procedure and the gastroenterology fellows performing the procedure.

Sample Size Based on a previous study measuring discomfort of patients undergoing colonoscopy we hypothesized that music can decrease the sedative/narcotic usage by 20 to 25 percent [25]. We expect a difference of 0.32mg/kg difference with a standard deviation of 0.69. Based on this, with a power of 90% and alpha of 0.05, we need 128 patients per group for a total of 384 patients. We plan to enroll 460 patients (over 18-years of age) to include a 20% dropout rate due to lack of compliance with headphones, inability to complete the exam, or failure to finish all accompanied documentation.

Recruitment Methods and Study Sites The study coordinator or investigators at The Brooklyn Hospital will approach all patients at the time of registration for colonoscopy. The coordinator will explain the study briefly and if agreeable will be given an iPad with a prerecorded video explaining the study in detail. After informed consent, patients will be randomized to either the control group (no music) or music group via a sealed envelope. A sealed envelope will delineate the particular group the patient will be randomized to. Once randomized, both groups will fill out a State Trait Anxiety Inventory (STAI) form to determine the baseline anxiety stress levels (Appendix A). This will be followed by a brief form (Appendix B) that will determine the type and number of procedures performed in the past. The forms will be administered in English, Spanish and Polish. Spanish and Polish translation will be provided using telephone medical translation services at The Brooklyn Hospital Center.

Data Collection and Storage Confidentiality of research data will be protected in accordance with the prevailing standards that apply to all clinical data. The binder with the data collection form and patient information will, as mentioned above, be locked in a filing cabinet in the GI endoscopy suit and will be reviewed only by the key study personnel. The patients' electronic health records, which contain the remainder of the patient data, are password protected. No personal identifying information will be used in any presentation or publication. The principal investigator and co-investigators will monitor study procedures to ensure confidentiality of data, safety and proper conduct of the study. Changes to the study will only occur after IRB amendment approval.

Risks and Benefits Utilizing headphones which can place a slight pressure around the ear, posing a very minimal risk. There is also a very rare possibility of hearing damage due to loud music being played on the headphones. To prevent this, the patient will adjust the music to his or her desired level with audible tones for both groups in the study prior to starting the music. There is a slight possibility of the loss of confidentiality, however this will be minimized by keeping all study related materials and data collection forms in a locked file cabinet as described above. Please refer to the confidentiality section of the protocol. Breaches of confidentiality, protocol deviations and any adverse events or other problems that may affect the safety of the subjects will be reported to the IRB in a timely fashion This study does not involve greater risk to the subjects than what is normally encountered during the performance of routine physical tests.

The benefit of the study is to demonstrate an overall improvement in sedation and patient satisfaction while decreasing the total amount of sedatives utilized.

Waiver of HIPAA Informed Consent This is a single blind prospective study that involves standard of care with human subjects. When not in use by the researchers, the data collection forms will be kept in a locked file cabinet located in Division of Gastroenterology and Hepatology, The Brooklyn Hospital Center, 240 Willoughby St., Maynard building, 2nd floor. Patient's data will be recorded in the computer and will be protected throughout the study in usual ways for IT security. The data collection form to be used is attached. All patient identifiers will be de-identified upon completion of data collection.

Resources and Budget The study is not funded and does not require extra lab tests, clinic visits, or supplies outside of standard clinical care. Therefore, these will not incur any additional costs for either the patients or the institution. There is no budget associated with this project as investigators will participate on a volunteer basis. There is no pay/stipend for study participants. Study personnel are limited to the participating gastroenterology, internal medicine, and research staff at the Brooklyn Hospital Center. No expenses will be incurred and nothing will be gained other than normal scholarly gains.

Conclusions Our results will improve patient satisfaction, reduce post-surgery complications and lessen the anxiety surrounding endoscopic procedures such as colonoscopies. It is our hope that improving our understanding of the role of music in regards to anxiety related colonoscopies, through a prospective, randomized, controlled research study, can help better facilitate patient care and outcomes and serve our population at the Brooklyn Hospital Center.

ELIGIBILITY:
Inclusion Criteria:

* Anyone scheduled for in-patient colonoscopy
* Must be able to speak English, Spanish, or Polish

Exclusion Criteria:

* Hearing impairment
* Mentally challenged
* Previous resection of the colon
* Currently using narcotics or sedative medications
* If patient is unwilling to use headphones after consenting

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include all individuals undergoing colonoscopies that consented to participating in the study. The study subjects will include the patients undergoing the procedure and the gastroenterology fellows performing the procedure.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-01-30 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Amount of sedation used | Duration of procedure
  Total dose of propofol will be calculated by the Anesthesiologist's team. The total dosage for each group will be compared using a t-test

SECONDARY OUTCOMES:
Anxiety levels and willingness to perform procedures | Duration of procedure
  Surveys will be used to assess anxiety levels and willingness to perform procedures. Contingency tables using Pearson's chi-squared test will be used to compare the two groups.
Effect of music in relation to level of trainee | Duration of procedure
  To assess the ordinal data with the year of the trainee using contingency tables and Pearson Chi-squared test

CONTACTS AND LOCATIONS:
Overall Officials: Krishna Gurram, MD, Principal Investigator — The Brooklyn Hospital Center; Daryl Ramai, MD, MScBR, Principal Investigator — The Brooklyn Hospital Center; Khoi Paul Dang-Ho, Principal Investigator — The Brooklyn Hospital Center; Madhavi Reddy, MD, Principal Investigator — The Brooklyn Hospital Center; Denzil Etienne, MD, Principal Investigator — The Brooklyn Hospital Center
Locations (1):
- The Brooklyn Hospital Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Froehlich F, Schwizer W, Thorens J, Kohler M, Gonvers JJ, Fried M. Conscious sedation for gastroscopy: patient tolerance and cardiorespiratory parameters. Gastroenterology. 1995 Mar;108(3):697-704. doi: 10.1016/0016-5085(95)90441-7. PMID 7875472
- [Background] Bini EJ, Firoozi B, Choung RJ, Ali EM, Osman M, Weinshel EH. Systematic evaluation of complications related to endoscopy in a training setting: A prospective 30-day outcomes study. Gastrointest Endosc. 2003 Jan;57(1):8-16. doi: 10.1067/mge.2003.15. PMID 12518123
- [Background] Qadeer MA, Rocio Lopez A, Dumot JA, Vargo JJ. Risk factors for hypoxemia during ambulatory gastrointestinal endoscopy in ASA I-II patients. Dig Dis Sci. 2009 May;54(5):1035-40. doi: 10.1007/s10620-008-0452-2. Epub 2008 Nov 12. PMID 19003534
- [Background] Sharma VK, Nguyen CC, Crowell MD, Lieberman DA, de Garmo P, Fleischer DE. A national study of cardiopulmonary unplanned events after GI endoscopy. Gastrointest Endosc. 2007 Jul;66(1):27-34. doi: 10.1016/j.gie.2006.12.040. PMID 17591470
- [Background] Clarke GA, Jacobson BC, Hammett RJ, Carr-Locke DL. The indications, utilization and safety of gastrointestinal endoscopy in an extremely elderly patient cohort. Endoscopy. 2001 Jul;33(7):580-4. doi: 10.1055/s-2001-15313. PMID 11473328
- [Background] Flegal KM, Carroll MD, Ogden CL, Curtin LR. Prevalence and trends in obesity among US adults, 1999-2008. JAMA. 2010 Jan 20;303(3):235-41. doi: 10.1001/jama.2009.2014. Epub 2010 Jan 13. PMID 20071471
- [Background] Bolwerk CA. Effects of relaxing music on state anxiety in myocardial infarction patients. Crit Care Nurs Q. 1990 Sep;13(2):63-72. doi: 10.1097/00002727-199009000-00009. No abstract available. PMID 2383784
- [Background] Byers JF, Smyth KA. Effect of a music intervention on noise annoyance, heart rate, and blood pressure in cardiac surgery patients. Am J Crit Care. 1997 May;6(3):183-91. PMID 9131197
- [Background] Colt HG, Powers A, Shanks TG. Effect of music on state anxiety scores in patients undergoing fiberoptic bronchoscopy. Chest. 1999 Sep;116(3):819-24. doi: 10.1378/chest.116.3.819. PMID 10492293
- [Background] Cunningham MF, Monson B, Bookbinder M. Introducing a music program in the perioperative area. AORN J. 1997 Oct;66(4):674-82. doi: 10.1016/s0001-2092(06)62920-7. PMID 9337469
- [Background] Guzzetta CE. Effects of relaxation and music therapy on patients in a coronary care unit with presumptive acute myocardial infarction. Heart Lung. 1989 Nov;18(6):609-16. PMID 2684920
- [Background] Sarkamo T, Tervaniemi M, Laitinen S, Forsblom A, Soinila S, Mikkonen M, Autti T, Silvennoinen HM, Erkkila J, Laine M, Peretz I, Hietanen M. Music listening enhances cognitive recovery and mood after middle cerebral artery stroke. Brain. 2008 Mar;131(Pt 3):866-76. doi: 10.1093/brain/awn013. PMID 18287122
- [Background] Sendelbach SE, Halm MA, Doran KA, Miller EH, Gaillard P. Effects of music therapy on physiological and psychological outcomes for patients undergoing cardiac surgery. J Cardiovasc Nurs. 2006 May-Jun;21(3):194-200. doi: 10.1097/00005082-200605000-00007. PMID 16699359
- [Background] Wang SM, Kulkarni L, Dolev J, Kain ZN. Music and preoperative anxiety: a randomized, controlled study. Anesth Analg. 2002 Jun;94(6):1489-94, table of contents. doi: 10.1097/00000539-200206000-00021. PMID 12032013
- [Background] White JM. Music therapy: an intervention to reduce anxiety in the myocardial infarction patient. Clin Nurse Spec. 1992 Summer;6(2):58-63. PMID 1617576
- [Background] El-Hassan H, McKeown K, Muller AF. Clinical trial: music reduces anxiety levels in patients attending for endoscopy. Aliment Pharmacol Ther. 2009 Oct;30(7):718-24. doi: 10.1111/j.1365-2036.2009.04091.x. Epub 2009 Jul 8. PMID 19604181
- [Background] Hayes A, Buffum M, Lanier E, Rodahl E, Sasso C. A music intervention to reduce anxiety prior to gastrointestinal procedures. Gastroenterol Nurs. 2003 Jul-Aug;26(4):145-9. doi: 10.1097/00001610-200307000-00002. PMID 12920428
- [Background] Kotwal MR, Rinchhen CZ, Ringe VV. Stress reduction through listening to Indian classical music during gastroscopy. Diagn Ther Endosc. 1998;4(4):191-7. doi: 10.1155/DTE.4.191. PMID 18493472
- [Background] Oddby-Muhrbeck E, Jakobsson J. Recall of music: a comparison between anaesthesia with propofol and isoflurane. Acta Anaesthesiol Scand. 1993 Jan;37(1):33-7. doi: 10.1111/j.1399-6576.1993.tb03594.x. PMID 8424291
- [Background] Ayoub CM, Rizk LB, Yaacoub CI, Gaal D, Kain ZN. Music and ambient operating room noise in patients undergoing spinal anesthesia. Anesth Analg. 2005 May;100(5):1316-1319. doi: 10.1213/01.ANE.0000153014.46893.9B. PMID 15845676
- [Background] Kim DW, Kil HY, White PF. The effect of noise on the bispectral index during propofol sedation. Anesth Analg. 2001 Nov;93(5):1170-3. doi: 10.1097/00000539-200111000-00022. PMID 11682389
- [Background] Koelsch S, Fuermetz J, Sack U, Bauer K, Hohenadel M, Wiegel M, Kaisers UX, Heinke W. Effects of Music Listening on Cortisol Levels and Propofol Consumption during Spinal Anesthesia. Front Psychol. 2011 Apr 5;2:58. doi: 10.3389/fpsyg.2011.00058. eCollection 2011. PMID 21716581
- [Background] Lee DW, Chan KW, Poon CM, Ko CW, Chan KH, Sin KS, Sze TS, Chan AC. Relaxation music decreases the dose of patient-controlled sedation during colonoscopy: a prospective randomized controlled trial. Gastrointest Endosc. 2002 Jan;55(1):33-6. doi: 10.1067/mge.2002.120387. PMID 11756911
- [Background] Zhang XW, Fan Y, Manyande A, Tian YK, Yin P. Effects of music on target-controlled infusion of propofol requirements during combined spinal-epidural anaesthesia. Anaesthesia. 2005 Oct;60(10):990-4. doi: 10.1111/j.1365-2044.2005.04299.x. PMID 16179044